CLINICAL TRIAL: NCT01376739
Title: Drug Use Investigation of Magnevist
Brief Title: Magnevist Post-marketing Surveillance in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Head Medical Development Japan, Bayer Yakuhin Co. LTD.
Other Study IDs: 15035; MAGNEVIST
Record Dates: First submitted 2011-06-08; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-06

CONDITIONS: Diagnostic Imaging
Keywords: Magnevist; MR angiography
MeSH Terms: interventions — Gadolinium DTPA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — Patients who will need to undergo contrast enhanced MR angiography with Magnevist (a dosage of more than 0.2 mg/kg)

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Magnevist at a dose of more than 0.2 ml/kg for MR angiography of peripheral vasculature with continuous imaging from the abdomen to the lower extremities. The objective of this study is to assess safety, especially in relation to renal dysfunction, and efficacy of using Magnevist in clinical practice. A total 2,000 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a dose of more than 0.2 mg/kg of Magnevist for MR angiography of peripheral vasculature with continuous imaging from the abdomen to the lower extremities

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who received Magnevist for MR angiography. The study is expected to collect data of 2,000 patients in approximately 150 hospitals in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 2051 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subjects who received Magnevist | After Magnevist administration, up to 3 years
Incidence of adverse drug reactions, especially Nephrogenic Systemic Fibrosis and Nephrogenic Fibrosing Dermopathy (NSF/NFD) in patients with reduced renal functions | After Magnevist administration, up to 3 years

SECONDARY OUTCOMES:
MRI image evaluation assessment by the four rank scales of 1 to 4: 1) sufficient extraction; 2) almost sufficient extraction; 3) not sufficient extraction; and 4) insufficient extraction | After Magnevist injection, up to 3 years
Incidence of adverse drug reactions in subpopulation with baseline data | At baseline and after Magnevist administration, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan